CLINICAL TRIAL: NCT04480099
Title: The Efficacy and Safety of Targeted Drug in Combination With Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP) in the Treatment of Newly Diagnosed Peripheral T-Cell Lymphoma
Brief Title: Targeted Drug Combined With CHOP in the Treatment of Newly Diagnosed Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director，Hematology Department, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-PTCL-1
Record Dates: First submitted 2020-07-19; First posted 2020-07-21 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma; Targeted therapy
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHOP (Active Comparator): Patients in this arm will receive conventional CHOP regimen for 6 cycles
  Interventions: Drug: CHOP
- CHOP+X (Experimental): Patients in this arm will receive targeted drug in combination with conventional CHOP regimen for 6 cycles, based on NGS results
  Interventions: Drug: CHOP+X

INTERVENTIONS:
Drug: CHOP — Cyclophosphamide 750mg/m2, ivgtt D1, doxorubicin 50mg/m2,ivgtt D1 Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 6 courses
  Arms: CHOP
Drug: CHOP+X — X: X(i.e. targeted drug) will decided by NGS results as following. Decitabine 10mg/m2 ivgtt D-5 to-1 if with TP53 gene muation. Azacitadine 100mg/day ivgtt D-7 to -1 if with TET2/KMT2D gene mutation. Chidamide 20mg/day po D1,4,8,11 if with CREBBP/EP300 gene mutation. Lenalidomide 25mg/day po D1-10 if without gene mutation above. X will be added from the second cycle CHOP:Cyclophosphamide 750mg/m2, ivgtt D1, doxorubicin 50mg/m2,ivgtt D1 Vincristine 1.4mg/m2（max 2mg）, ivgtt D1 Prednisone 60mg/m2 （max 100mg）,PO,D1-D5 every 21 days for total 6 courses
  Arms: CHOP+X

SUMMARY:
This prospective，multi-center，open-label, controlled study will evaluate the efficacy and safety of targeted drug in combination with CHOP in treatment of newly diagnosed peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL）is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for ~10%. Patients with PTCL still have poor treatment response and prognosis under conventional CHOP regimen. There is no standard of care for those patients. Targeted drugs are warranted in this group of patients to improve survival. This prospective，multi-center，open-label, controlled study will evaluate the efficacy and safety of targeted drug in combination with CHOP in treatment of newly diagnosed peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed peripheral T-cell lymphoma based on 2016 WHO classification with enough tumor sample for NGS
* Treatment naive
* Age ≥ 18 years
* Must has measurable lesion in CT or PET-CT prior to treatment
* ECOG 0,1,2
* Informed consented

Exclusion Criteria:

* ALCL,ALK positive, NK/T-cell leukemia, adult T-cell lymphoma/leukemia, T-LGL
* Has accepted localized or systemic anti-lymphoma treatment
* Has accepted autologous Stem cell transplantation before
* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix prior to study treatment
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Primary CNS lymphoma
* Left EF≤ 50%
* Lab at enrollment (Unless caused by lymphoma): Neutrophile<1.5*10^9/ L ;Platelet<50*10^9/L; ALT or AST >2*ULN; Creatinine>1.5*ULN
* Other uncontrollable medical condition that may that may interfere the participation of the study
* Not able to comply to the protocol for mental or other unknown reasons
* Patients with mentally disorders or other reasons unable to fully comply with the study protocol
* Pregnant or lactation
* HIV infection
* HBV-DNA or HCV-RNA positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria

SECONDARY OUTCOMES:
Overall response rate | At the end of Cycle 6 (each cycle is 21 days)
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria
Progression free survival | Baseline up to data cut-off (up to approximately 4 years)
  Progression-free survival was defined as the time from the date of diagnosis until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
Treatment related mortality | Baseline up to data cut-off (up to approximately 4 years)
  Percentage of death related with treatment on the basis of investigator assessments
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC QLQ-C30) Domain Scores | Baseline (pre-dose [Hour 0] on Cycle1 Day1), Cycle3 Day 1, end of treatment (up to Month 6), every 3 months 1st year, every 6 months 2nd year, and 12 months thereafter up to data cut-off, up to approximately 4 years (cycle length = 21 days)
  The EORTC QLQ-C30 is a health-related quality of life questionnaire. A higher score indicates better quality of life, with changes of 5 to 10 points considered to be a minimally important difference to participants.

OTHER OUTCOMES:
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  CfDNA in peripheral blood assessed by local lab
Exploratory biomarker analysis | Baseline up to data cut-off (up to approximately 4 years)
  Exploratory biomarker to predict treatment response and survival

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Department of Hematology, Peking University Third Hospital, Beijing, China, Beijing
  - Department of Hematology, West China Hospital, Sichuan University, Chengdu, Sichuan, China, Chengdu
  - Department of Hematology, Fujian Institute of Hematology, Fujian Provincial Key Laboratory on Hematology, Union Hospital, Fujian Institute of Hematology, Fuzhou, China, Fuzhou
  - Department of Hematology, Shandong Provincial Hospital Affiliated to Shandong University, Jinan, China, Shandong
  - Shanghai Ruijin Hospital, Shanghai
  - Department of Hematology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China, Wuhan
  - Department of Hematology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China, Wuhan

REFERENCES:
- [Derived] Cai MC, Cheng S, Jing HM, Liu Y, Cui GH, Niu T, Shen JZ, Huang L, Wang X, Huang YH, Wang L, Xu PP, Zhao WL. Targeted agents plus CHOP compared with CHOP as the first-line treatment for newly diagnosed patients with peripheral T-cell lymphoma (GUIDANCE-03): an open-label, multicentre phase 2 clinical trial. Lancet Reg Health West Pac. 2024 Jul 29;50:101160. doi: 10.1016/j.lanwpc.2024.101160. eCollection 2024 Sep. PMID 39175480